CLINICAL TRIAL: NCT00253422
Title: A Partially Blind Phase III Randomised Trial of Faslodex +/- Concomitant Arimidex Compared With Exemestane in Post-menopausal Women With ER+ or PR+ Locally Advanced/Metastatic Breast Cancer Following Progression on Non-steroidal AIs
Brief Title: Study of Faslodex +/- Concomitant Arimidex v Exemestane Following Progression on Non-steroidal Aromatase Inhibitors
Acronym: SoFEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000448616; ICR-CTSU-SOFEA (Other: ICR-CTSU); ISRCTN44195747 (Other: ISRCTN); MREC-03677 (Other: REC); 2004-000093-30 (EudraCT Number)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Arimidex vs Arimidex-placebo component is double-blinded. Faslodex is not blinded Exemestane is not blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Faslodex + placebo (Active Comparator): Arimidex/placebo comparator is blinded Faslodex (fulvestrant) IM on day 1,15,29 and monthly thereafter Placebo orally once a day
  Interventions: Drug: Anastrozole; Drug: Fulvestrant
- Faslodex + Arimidex (Active Comparator): Arimidex/placebo comparator is blinded Faslodex (fulvestrant) IM on day 1,15,29 and monthly thereafter Arimidex (anastrozole) orally once a day
  Interventions: Drug: Anastrozole; Drug: Fulvestrant
- Exemestane (Active Comparator): exemestane orally once a day
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Anastrozole — This may be Anastrazole OR a placebo
  Other Names: Arimidex (or placebo)
  Arms: Faslodex + Arimidex; Faslodex + placebo
Drug: Exemestane
  Arms: Exemestane
Drug: Fulvestrant
  Other Names: Faslodex
  Arms: Faslodex + Arimidex; Faslodex + placebo

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant, anastrozole, or exemestane may fight breast cancer by blocking the use of estrogen by the tumor cells or by lowering the amount of estrogen the body makes. It is not yet known whether giving fulvestrant together with anastrozole is more effective than giving fulvestrant together with a placebo or exemestane alone in treating breast cancer.

PURPOSE: This randomized phase III trial is studying fulvestrant and anastrozole to see how well they work compared to fulvestrant and a placebo or exemestane alone in treating postmenopausal women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of postmenopausal women with estrogen receptor- and/or progesterone receptor-positive, locally advanced or metastatic breast cancer that relapsed or progressed during prior treatment with nonsteroidal aromatase inhibitors treated with fulvestrant with vs without anastrozole vs exemestane alone.

Secondary

* Compare the objective complete response (CR) and partial response (PR) rate and duration of response in patients treated with these regimens.
* Compare the clinical benefit (i.e., 6-month CR, PR, and stable disease) rate and duration of clinical benefit in patients treated with these regimens.
* Compare time to treatment failure in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.

OUTLINE: This is a randomized, partially double-blind and placebo-controlled, multicenter study. Patients are stratified according to the setting in which prior nonsteroidal aromatase-inhibitor therapy was given (adjuvant therapy vs first-line therapy) and participating center. Patients are randomized to 1 of 3 treatment arms.

* Arm I (fulvestrant and anastrozole): Patients receive fulvestrant intramuscularly (IM) on days 1, 15, and 29 and then once monthly. Patients receive oral anastrozole once daily.
* Arm II (fulvestrant and placebo): Patients receive fulvestrant as in arm I and oral placebo once daily.
* Arm III (exemestane alone): Patients receive oral exemestane once daily. In all arms, treatment repeats every month in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 750 patients (250 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Locally advanced or metastatic disease
* Metastatic disease must be measurable or evaluable

  * Patients with bone only metastases are eligible provided there is an evaluable site of bone metastasis that can be followed by x-ray, MRI, or CT scan
* Relapsed or progressed during prior treatment with single-agent nonsteroidal aromatase inhibitor (NSAI)*, meeting either of the following criteria:

  * NSAI given as adjuvant therapy that lasted ≥ 12 months
  * Achieved an objective complete response, partial response, or stable disease that lasted ≥ 6 months after prior first-line therapy with NSAI for locally advanced or metastatic disease

    * Chemotherapy as part of the first-line therapy given before initiation of NSAI allowed NOTE: *Patients are required to continue to take NSAI until beginning of study treatment.
* No rapidly progressive visceral disease (i.e., lymphangitis carcinomatosa or diffuse hepatic involvement)
* Hormone receptor status:

  * Estrogen receptor (ER) and/or progesterone receptor positive tumor
  * No ER-unknown disease

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Postmenopausal, as defined by 1 of the following criteria:

  * Age 60 and over
  * Age 45 to 59 AND ≥ 12 months since last menstrual period with no prior hysterectomy
  * Any age with prior bilateral oophorectomy

Performance status

* WHO 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

  * No thrombocytopenia
* Hemoglobin ≥ 10 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN (unless due to bone metastases)
* No liver disease

Renal

* Creatinine < 1.97 mg/dL

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* Prior neoadjuvant or adjuvant chemotherapy allowed

Endocrine therapy

* See Disease Characteristics
* Prior tamoxifen as neoadjuvant or adjuvant therapy allowed
* No systemic corticosteroids that lasted > 15 days within the past 4 weeks

Other

* More than 4 weeks since prior investigational drugs
* Concurrent bisphosphonates for bone metastases allowed provided bisphosphonate therapy has been established for ≥ 6 months

  * Concurrent initiation of bisphosphonate allowed provided patient has soft tissue or visceral metastases as the measurable or evaluable target lesion
* No concurrent anticoagulant therapy
* No concurrent unlicensed noncancer investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2004-03-26 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen RD Johnston, MD,PhD,FRCP, Study Chair — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Marsden - London, London, England
  - Institute Of Cancer Research, Sutton, England

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, together with a data dictionary defining each field in the set, will be made available to other researchers on request, subject to the approval of a formal data access request in accordance with the ICR-CTSU data and sample access policy. Trial documentation including the protocol are available on request by contacting Formal requests for data sharing are considered in line with ICR-CTSU procedures. Requests are via a standard proforma describing the nature of the proposed research and extent of data requirements. Contact sofea-icrctsu@icr.ac.uk or visit the link below for further information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available to researchers following the formal review and approval of a data access request in accordance with the ICR-CTSU data and sample access policy.
Access Criteria: Completion and approval of a data access request form as stated above
URL: https://www.icr.ac.uk/our-research/centres-and-collaborations/centres-at-the-icr/clinical-trials-and-statistics-unit/working-with-us/data-sharing

REFERENCES:
- [Result] Johnston SR, Kilburn LS, Ellis P, Dodwell D, Cameron D, Hayward L, Im YH, Braybrooke JP, Brunt AM, Cheung KL, Jyothirmayi R, Robinson A, Wardley AM, Wheatley D, Howell A, Coombes G, Sergenson N, Sin HJ, Folkerd E, Dowsett M, Bliss JM; SoFEA investigators. Fulvestrant plus anastrozole or placebo versus exemestane alone after progression on non-steroidal aromatase inhibitors in postmenopausal patients with hormone-receptor-positive locally advanced or metastatic breast cancer (SoFEA): a composite, multicentre, phase 3 randomised trial. Lancet Oncol. 2013 Sep;14(10):989-98. doi: 10.1016/S1470-2045(13)70322-X. Epub 2013 Jul 29. PMID 23902874
- [Derived] Fribbens C, O'Leary B, Kilburn L, Hrebien S, Garcia-Murillas I, Beaney M, Cristofanilli M, Andre F, Loi S, Loibl S, Jiang J, Bartlett CH, Koehler M, Dowsett M, Bliss JM, Johnston SR, Turner NC. Plasma ESR1 Mutations and the Treatment of Estrogen Receptor-Positive Advanced Breast Cancer. J Clin Oncol. 2016 Sep 1;34(25):2961-8. doi: 10.1200/JCO.2016.67.3061. Epub 2016 Jun 6. PMID 27269946
- See also: Clinical trial summary from ICR website — https://www.icr.ac.uk/research-and-discoveries/centres-and-strategic-collaborations/clinical-trials-and-statistics-unit-icr-ctsu/detail/sofea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 26 March 2004 and 6 August 2010 from 82 hospitals in the UK.
Pre-assignment Details: Prior to randomisation patients were assessed for medical history and had a clinical examination, haematology and biochemistry and tumour staging to assess eligibility.
Groups:
- Exemestane: exemestane orally once a day
  Exemestane
Period: Overall Study
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Started | 226 | 233 | 239
Completed | 226 | 233 | 238
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Faslodex + Placebo: Arimidex/placebo comparator is blinded Faslodex (fulvestrant) IM on day 1,15,29 and monthly thereafter Placebo orally once a day
  Anastrozole: This may be Anastrazole OR a placebo
  Fulvestrant
- Faslodex + Arimidex: Arimidex/placebo comparator is blinded Faslodex (fulvestrant) IM on day 1,15,29 and monthly thereafter Arimidex (anastrozole) orally once a day
  Anastrozole: This may be Anastrazole OR a placebo
  Fulvestrant
- Total: Total of all reporting groups
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane | Total
Number analyzed (Participants) | 226 | 233 | 239 | 698
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.2 [57.0 to 73.6] | 64.1 [57.6 to 72.3] | 66.1 [59.2 to 75.3] | 64.7 [58.0 to 73.5]
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 17 | 21 | 7 | 45
  50 to 64 years | 102 | 104 | 100 | 306
  65 to 74 years | 61 | 65 | 70 | 196
  >=75 years | 46 | 43 | 62 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 233 | 239 | 698
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 226 | 233 | 239 | 698
Hormone Receptor Status of primary disease [Count of Participants; unit: Participants]
  ER+ve PR+ve | 121 | 111 | 123 | 355
  ER+ve PR -ve | 31 | 38 | 22 | 91
  ER+ve PR unknown | 71 | 83 | 91 | 245
  ER-ve/unknown PR+ve | 0 | 1 | 2 | 3
  ER unknown PR unknown | 2 | 0 | 1 | 3
  ER-ve PR-ve | 1 | 0 | 0 | 1
HER2 Status of primary disease [Count of Participants; unit: Participants]
  HER2 +ve | 14 | 15 | 15 | 44
  HER2 -ve | 136 | 117 | 134 | 387
  HER2 unknown | 76 | 101 | 90 | 267
Time from primary diagnosis to first relapse [Median (Inter-Quartile Range); unit: years] | 5.1 [2.3 to 9.6] | 5.0 [2.0 to 10.0] | 5.2 [1.9 to 10.3] | 5.1 [2.1 to 10.0]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: defined as time from randomisation to progression of existing disease, new sites of disease, second primary cancer if change in systemic treatment was necessary, or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessed up to 190 months
Population: Intention to treat (ITT). This population contains all people randomised into the study (regardless of whether they were later found to be ineligible, a protocol deviator, given the wrong treatment allocation, never treated etc.). Comparisons are made by randomised treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 226 | 233 | 239
Months | 4.8 [3.5 to 5.6] | 4.1 [3.2 to 5.3] | 3.5 [3.0 to 4.9]
Statistical Analysis 1: Comparison: Faslodex + Placebo vs Faslodex + Arimidex; Test type: Superiority; p = 0.76, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.86 to 1.24]
Statistical Analysis 2: Comparison: Faslodex + Placebo vs Exemestane; Test type: Superiority; p = 1.00, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.83 to 1.20]

2. Secondary Outcome: Objective Response Rate
Description: The proportion of patients identified as having a complete response (CR) or partial response (PR) at any time whilst on study treatment. Response is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as either disappearance of all lesions or a >=30% decrease in the sum of the longest diameter of target lesions with no progressing non-target lesions and no new lesions. Objective Response (OR) = CR + PR
Time Frame: From start of treatment, every 3 months to treatment discontinuation and/or up to 190 months
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- Faslodex + Placebo: Arimidex/placebo comparator is blinded Faslodex (fulvestrant) IM on day 1,15,29 and monthly thereafter Arimidex (anastrozole) or placebo orally once a day
  Anastrozole: This may be Anastrazole OR a placebo
  Fulvestrant
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 226 | 233 | 239
Participants | 16 | 17 | 10
Statistical Analysis 1: Comparison: Faslodex + Placebo vs Faslodex + Arimidex; Test type: Superiority; p = 0.99, Chi-squared
Statistical Analysis 2: Comparison: Faslodex + Placebo vs Exemestane; Test type: Superiority; p = 0.12, Chi-squared

3. Secondary Outcome: Duration of Response
Description: time from first assessment of response to progression or death. Response is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as either disappearance of all lesions or a >=30% decrease in the sum of the longest diameter of target lesions with no progressing non-target lesions and no new lesions. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessed up to 190 months
Population: The number of patients that had an objective response
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 16 | 17 | 10
Months | 10.2 [2.6 to 18.4] | 8.7 [3.0 to 12.2] | 12.8 [6.2 to 33.4]

4. Secondary Outcome: Clinical Benefit Rate
Description: Complete or partial response or stable disease for at least six months prior to progression. Response is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as either disappearance of all lesions or a >=30% decrease in the sum of the longest diameter of target lesions with no progressing non-target lesions and no new lesions. Stable disease is neither responding or progressing. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessed up to 190 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 226 | 233 | 239
Participants | 55 | 66 | 57
Statistical Analysis 1: Comparison: Faslodex + Placebo vs Faslodex + Arimidex; Test type: Superiority; p = 0.33, Chi-squared
Statistical Analysis 2: Comparison: Faslodex + Placebo vs Exemestane; Test type: Superiority; p = 0.94, Chi-squared

5. Secondary Outcome: Duration of Clinical Benefit
Description: Time from first assessment of clinical benefit to progression or death. Response is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as either disappearance of all lesions or a >=30% decrease in the sum of the longest diameter of target lesions with no progressing non-target lesions and no new lesions. Stable disease is neither responding or progressing. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Clinical benefit = (CR+PR)+(SD>=6months).
Time Frame: Assessed up to 190 months
Population: The number of patients that had clinical benefit, defined as complete or partial response, or stable disease for at least 6 months prior to progression.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 55 | 66 | 57
months | 11.2 [8.2 to 16.9] | 11.5 [8.0 to 16.3] | 12.2 [8.9 to 23.8]

6. Secondary Outcome: Time to Treatment Failure
Description: Time from randomisation to discontinuation of protocol treatment for any reason, or progression of disease
Time Frame: To discontinuation of protocol treatment for any reason, or progression of disease assessed up to 190 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 226 | 233 | 239
Months | 3.8 [3.1 to 5.4] | 3.9 [3.0 to 4.7] | 3.4 [3.1 to 4.5]
Statistical Analysis 1: Comparison: Faslodex + Placebo vs Faslodex + Arimidex; Test type: Superiority; p = 0.95, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.21] — HR less than 1 favour Faslodex + Arimidex
Statistical Analysis 2: Comparison: Faslodex + Placebo vs Exemestane; Test type: Superiority; p = 0.66, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.87 to 1.25] — HR less than 1 favours Faslodex + placebo

7. Secondary Outcome: Overall Survival
Description: Time from randomisation until death from any cause.
Time Frame: To death assessed up to 190 months.
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 226 | 233 | 239
Months | 20.1 [17.8 to 23.3] | 20.2 [17.0 to 22.6] | 22.5 [20.1 to 24.6]
Statistical Analysis 1: Comparison: Faslodex + Placebo vs Faslodex + Arimidex; Test type: Superiority; p = 0.91, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19] — HR less than 1 favours Faslodex + Arimidex
Statistical Analysis 2: Comparison: Faslodex + Placebo vs Exemestane; Test type: Superiority; p = 0.31, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.91 to 1.32] — HR less than 1 favours Faslodex + Placebo

8. Secondary Outcome: Tolerability of Treatment
Description: To evaluate the overall safety and tolerability. The number of patients experiencing at least one adverse event. Refer to adverse event section for more details.
Time Frame: From start of treatment to discontinuation of treatment/progression assessed up to 190 months
Population: Number of patients that received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
Number analyzed (Participants) | 225 | 231 | 237
Participants | 221 | 227 | 230

ADVERSE EVENTS:
Time Frame: Collected from the date each patient commenced treatment. AEs were collected every month for the first six months of the protocol and then every three months until disease progression/treatment discontinuation (assessed up to 190 months).
Description: All events were graded according to CTCAE V3.0.
  For (S)AEs the analysis population was "as treated", i.e. all patients receiving at least one dose of treatment. For all cause mortality the analysis population is ITT.
Arm/Group | Faslodex + Placebo | Faslodex + Arimidex | Exemestane
All-Cause Mortality (participants affected / at risk) | 221/226 | 225/233 | 227/239
Serious Adverse Events (participants affected / at risk) | 31/225 | 39/231 | 37/237
Other Adverse Events (participants affected / at risk) | 221/225 | 227/231 | 230/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faslodex + Placebo (N=225) | Faslodex + Arimidex (N=231) | Exemestane (N=237)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1
Lymphangitis (Blood and lymphatic system disorders) | 1 | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac operation (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 3 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Abdominal abscess (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 2 | 4 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2
Chest pain (General disorders) | 1 | 0 | 3
Fatigue (General disorders) | 3 | 0 | 1
Lethargy (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 1
Swelling (General disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 3
Lung abscess (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 3
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Infections and infestations) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intramedullary rod insertion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Haematemesis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1
Penetrating aortic ulcer (Vascular disorders) | 0 | 0 | 1
Presyncope (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faslodex + Placebo (N=225) | Faslodex + Arimidex (N=231) | Exemestane (N=237)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (71) | 25 (59) | 32 (68)
Arthralgia (Musculoskeletal and connective tissue disorders) | 98 (304) | 97 (314) | 110 (318)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (37) | 17 (23) | 21 (28)
Bone Pain (Musculoskeletal and connective tissue disorders) | 12 (18) | 19 (34) | 20 (32)
Constipation (Gastrointestinal disorders) | 57 (124) | 64 (172) | 57 (135)
cough (Respiratory, thoracic and mediastinal disorders) | 19 (39) | 7 (8) | 16 (29)
decreased appetite (Metabolism and nutrition disorders) | 67 (145) | 72 (121) | 68 (127)
diarrhoea (Gastrointestinal disorders) | 53 (105) | 39 (68) | 49 (71)
Dizziness (Nervous system disorders) | 10 (10) | 12 (19) | 15 (17)
Dyspepsia (Gastrointestinal disorders) | 59 (150) | 51 (105) | 70 (122)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (61) | 16 (23) | 25 (45)
Headache (Nervous system disorders) | 65 (153) | 51 (119) | 51 (114)
Hot Flush (Reproductive system and breast disorders) | 81 (282) | 86 (278) | 79 (215)
Insomnia (Psychiatric disorders) | 64 (192) | 76 (207) | 70 (204)
Lethargy (General disorders) | 145 (436) | 149 (432) | 133 (386)
Lower respiratory tract infection (Infections and infestations) | 16 (19) | 17 (23) | 13 (14)
Mood altered (Psychiatric disorders) | 59 (157) | 55 (122) | 59 (113)
Mucosal Inflammation (General disorders) | 23 (57) | 15 (20) | 16 (21)
pain (General disorders) | 16 (27) | 5 (5) | 10 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (11) | 15 (29) | 14 (23)
Urinary tract infection (Infections and infestations) | 14 (17) | 8 (10) | 7 (8)
Vomiting (Gastrointestinal disorders) | 101 (224) | 81 (154) | 91 (147)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between principal investigators and the Sponsor (or its agents) that restricts the PIs rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-06-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT00253422/Prot_SAP_000.pdf